CLINICAL TRIAL: NCT01399671
Title: Clinical Randomized Trial to Evaluate the Efficacy of Vestibular Stimulation as Coadjuvant Therapy in Major Depression
Brief Title: Study of the Effectiveness of Vestibular Stimulation as a Coadjuvant Treatment in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuerza Aérea de Chile (Other Government)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Ana Maria Soza Ried, Dr, Fuerza Aérea de Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SA10I220044
Record Dates: First submitted 2011-07-12; First posted 2011-07-22 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2011-03

CONDITIONS: Depression; Major Depression; Vestibular Disorders
Keywords: depression; vestibular
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: vestibular stimulation — vestibular stimulation

SUMMARY:
Major depression is characterized by vestibular anomalies. The investigators hypothesized that vestibular stimulation will improve depression symptoms in major depression patients.

ELIGIBILITY:
Inclusion Criteria:

* major depression patients,
* actual Hamilton score > 14

Exclusion Criteria:

* pregnant,
* neurological disorders,
* epilepsy,
* bipolar disorder,
* schizophrenia,
* anorexia,
* bulimia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Hamilton depression rating score | 1 month after the treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Soza, MD, Principal Investigator — Fuerza Aerea de Chile
Locations (1):
- Centro de Medicina Aeroespacial, Santiago, Santiago Metropolitan, Chile